CLINICAL TRIAL: NCT06590519
Title: The Effectiveness of Date Seed Extract in Controlling Diabetes and Reducing Cardiovascular Risk in Patients With Type 2 Diabetes in Riyadh, Saudi Arabia
Brief Title: Date Seed Extract Effectiveness in Controlling Diabetes and Cardiovascular Risk in T2DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Maha Abdulrahman Aldaham, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UPM-PhD MAHA ALDAHAM
Record Dates: First submitted 2024-08-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
Who Masked: Participant
Masking Description: Single (Participants)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Date Seed Capsule (Other): The intervention group will receive a capsule of date-seed powder. Each person should consume 5 grams (two capsules of date-seed powder) twice daily after meals for three months. Assessments are carried out at the beginning of the study, one month and two months after the intervention (Chan et al., 2013). Participants will be contacted twice a week to ensure that they are adhering to the rules, maintaining their physical activity and clarifying any questions about taking supplements.
  Interventions: Other: Date Seed Extract
- Control group: No Intervention (No Intervention): The control group will not receive any capsule ot treatment.

INTERVENTIONS:
Other: Date Seed Extract — Intervention group participants will undergo a three-month intervention program. The Health Belief Model (HBM) will be the underlying theory to facilitate behaviour change.
  The intervention group will receive a capsule of date-seed-powder. Each person should consume 5 grams (two capsules of date-seed powder)twice daily after meals for three months.
  Assessments are carried out at the beginning of the study, one month and two months after the intervention on the effect of date-seed on glycaemic control,risk of cardiovascular, physical activity, daytime sleepiness and anthropometric measurements. Participants will be contacted twice a week to ensure that they are adhering to the rules.
  Other Names: Intervention group
  Arms: Date Seed Capsule

SUMMARY:
Globally, chronic noncommunicable diseases rank as the leading cause of morbidity and mortality. Diabetes is reaching high epidemic proportions across the globe. The prevalence of diabetes is increasing in Saudi Arabia, with diabetes affecting 14.1% of the population across all age groups and 28% of those over the age of 30. Date seed intake is one of the best-studied patterns. Previous studies findinds showed that the phenolic compounds in date seeds have blood sugar-lowering properties. There is a lack of data on how date seed diets may affect glycaemia control and cardiovascular risk among Saudi Arabian patients with T2DM. Therefore, randomised controlled trials (RCTs) will be conducted to assess the effects of date seeds on glycaemic control and cardiovascular risk among diabetes patients.

DETAILED DESCRIPTION:
A randomized controlled trial study will be conducted among adults with Type 2 diabetes who referred to the diabetes center to optimise dietary intervention for diabetes control in King Fahad Medical City (KFMC), Riyadh, Saudi Arabia. A total of 160 participants (80 participants for each group) will be select using simple random sampling.

The intervention group will receive a capsule of date-seed powder, while the control group will not receive any capsule. Each person should consume 5 grams (two capsules of date-seed powder) twice daily after meals for three months. Assessments are carried out at the beginning of the study, one month and two months after the intervention (Chan et al., 2013). Participants will be contacted twice a week to ensure that they are adhering to the rules, maintaining their physical activity and clarifying any questions about taking supplements. A checklist is also provided to all participants to monitor their adherence. Participants who fail to take more than 10% of the packs will be excluded from the study.

For the preparation of date seeds (Sukkari), firstly the desired concentrations of date seed powder for the different versions of Sukkari are determined. Secondly, the amount of date seed powder required for each concentration is calculated based on the total volume of the product. Then, separate containers are prepared for each version of Sukkari. A grinder is used to extract the bioactive substances from the date seeds and prepare the powder. First, the date seeds are washed and dried. Then we use a grinder and grind them into powder. Finally, gelatin capsules will be filled with date kernel powder, and then packed in identical containers.

The data will be collected from the intervention and control group before the intervention, one month after the intervention and two months follow-up after the intervention data collection through a self-administered questionnaire. The questionnaire will be consisted of eight sections aimed at obtaining information on socio-demographic data, lifestyle characteristics and clinical parameters of the study participants. Accordingly, dietary data and physical measurements, including anthropometric measurements, blood pressure and biochemical parameters, will be collected. Data will be analyzed by using the software Statistical Package for Social Sciences (SPSS) version 26.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old and above.
* Diagnosis of Type 2 diabetes.
* Receiving and monitoring diabetes care from diabetes center.
* With stable HbA1c less than 10% (no episode of hypoglycaemia, no hospitalisation, no change in type or dosage of medication use for at least 6 months).

Exclusion Criteria:

* Pregnant or lactating women.
* Diagnosis of cardiac failure or/and severe renal disease, with physical or mental disability, neurological or cognitive impairment.
* Participant with severely impaired vision, hearing, or speech.
* Participants who have known allergy to dates products.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Glucose Levels | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post intervention)]
  Fasting plasma glucose and Random blood glucose will be measured using a spectrophotometer. The normal range of the Fasting plasma glucose is (5.6 - 6.9 mmol/l) and for Random blood glucose is (7.8-11.0 mmol/l).
Change in cholesterol Levels | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post intervention)]
  Total cholesterol includes both High density lipoprotein cholesterol (HDL) and Low density lipoprotein cholesterol (LDL) will be measured using a spectrophotometer. The normal range of the total cholesterol is (≤ 5.2 mmol/l). While the normal range of LDL-cholesterol is (˂ 2.6 mmol/l) and HDL-cholesterol is (˃ 1.3 mmol/l)
Change in Blood Pressure | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post intervention)]
  Blood pressure will be measured using sphygmomanometer. Normal blood pressure is usually considered to be between 120/80 mmHg.

SECONDARY OUTCOMES:
Change the Body mass index (BMI) | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post intervention)]
  The Body mass index (BMI) will be report in kg/m^2 by using the following formula (BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared). Body weight will be measured using Omron HBF 375 to the nearest 0.1 kg. SECA body meter 206 will be employed to measure their heights to the nearest 0.1 cm. Body mass index (BMI) will be classified into (underweight, normal weight, overweight, and obesity). If the BMI is less than 18.5, it falls within the underweight range. If the BMI is 18.5 to <25, it falls within the healthy weight range. If the BMI is 25.0 to <30, it falls within the overweight range. If the BMI is 30.0 or higher, it falls within the obesity range.
Change in Change in physical activity | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post intervention)]
  Physical activity practice will be measured using international physical activity questionnaire (IPAQ). Time spent on all physical activity types will be summed to obtain each physical activity type's time spent per week. Frequency, duration, and intensity for each physical activity type were coded into metabolic equivalent (MET) tables. The total MET per week for all physical activities was calculated by multiplying the duration (minutes) of activity per week by its corresponding METs and summing for each physical activity type. Sufficient MET was defined as ≥600 METs per week.
Change in daytime sleepiness | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post intervention)]
  Participants' daytime sleepiness will be assessed using the Epworth Sleepiness Scale (ESS). Participants will be asked to rate their chances of dozing during certain daily activities using ratings range from 0 (never doze) to 3 (high chance of dozing). Scores range from 0 to 24. An ESS score greater than 10 indicates excessive daytime sleepiness.
Change in dietary intakes | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post intervention)]
  The 24-hour dietary recall will be used at baseline and at the end of the study to assess participants' dietary intake on two non-consecutive days (one usual day and one weekend day).

CONTACTS AND LOCATIONS:
Overall Officials: Zuriati Ibrahim, PhD, Principal Investigator — UniversitI Putra Malaysia (UPM), 43400 Serdang, Selangor, Malaysia
Locations (1):
- Dr Zuriati Ibrahim, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No